CLINICAL TRIAL: NCT01243593
Title: Transversus Abdominis Plane Block in Children Undergoing Open Pyeloplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000019942
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia
Keywords: pediatrics; anesthesia; pyeloplasty; Transversus Abdominis Plane Block; Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Procedure: Transversus Abdominis Plane Block
- Control Group (Active Comparator)
  Interventions: Procedure: Standard Anesthesia

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — A block needle will be advanced in a medial to lateral direction until the tip is visualized in the transversus abdominis plane. After negative aspiration 0.4 ml/kg of bupivacaine 0.25% with 1:200 000 epinephrine will be injected. The total dose of bupivacaine will not exceed 2 mg/kg and the total volume will not be more than 20 ml.
  Arms: Treatment Group
Procedure: Standard Anesthesia — Local field infiltration with bupivacaine 0.25% with 1:200 000 epinephrine 0.4 ml/kg before skin incision.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of transversus abdominis plane (TAP) block in reducing postoperative opioid requirements and pain after open pyeloplasty surgery in children.

DETAILED DESCRIPTION:
Primary open pyeloplasty is a common elective surgical procedure at The Hospital for Sick Children. All children are given fentanyl plus local anesthetic wound infiltration for intraoperative analgesia. A retrospective audit demonstrated that 63% of children required additional opioid treatment in the early recovery period following surgery. Concern exists regarding potential side effects of opioids including nausea or vomiting, respiratory depression, pruritus, over-sedation and delayed transition to oral intake. More importantly, children may under-report their pain or pain may not be recognized by medical staff leading to inadequate provision of analgesia. This suggests that the use of a regional technique, such as a TAP block, may benefit children undergoing open pyeloplasty.

The ultrasound guided TAP block introduces a local anaesthetic to the transversus abdominis plane which is one of three muscle layers in the abdominal wall. This results in a block of the nerves leading to the abdominal wall thereby reducing pain sensations.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification score 1-3
* age 1 month to 6 years inclusive

Exclusion Criteria:

* children undergoing an additional surgical procedure at an anatomical location not covered by a unilateral TAP block during the same anesthetic
* children in whom a TAP block is contraindicated, i.e. surgical scar or distorted anatomy at the site of injection
* postoperative admission to the intensive care unit
* children with a known allergy to bupivacaine
* children with a history of chronic abdominal pain requiring opioid analgesics
* children with known renal insufficiency
* children with known impaired hepatic function
* children with known impaired cardiac function
* children known hypersensitivity to sodium metabisulfite

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lorenzo AJ, Lynch J, Matava C, El-Beheiry H, Hayes J. Ultrasound guided transversus abdominis plane vs surgeon administered intraoperative regional field infiltration with bupivacaine for early postoperative pain control in children undergoing open pyeloplasty. J Urol. 2014 Jul;192(1):207-13. doi: 10.1016/j.juro.2014.01.026. Epub 2014 Feb 8. PMID 24518763

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 16 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.7 (0.2) | 1 (0.3) | 0.85 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 12 | 7 | 19
Weight [Mean (Standard Deviation); unit: kg] | 8.4 (0.62) | 9.2 (0.92) | 8.7 (3)

OUTCOME MEASURES:

1. Primary Outcome: Requirement for Morphine Post-surgery.
Description: The primary outcome measure will be the count and percentage of children who require morphine in the recovery room.
Time Frame: Time in recovery room, approximately 60-90 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 16
Participants | 13 | 6

2. Secondary Outcome: Total Amount of Morphine (mg/kg) Administered in the Recovery Room.
Description: Patients will receive intravenous morphine 0.05 mg/kg if the FLACC is ≥ 3/10 (equivalent to mild-to-moderate pain). Morphine may be given at 10 minute intervals as per standard protocol until the FLACC score is < 3/10, or the child declines additional pain medicine when offered.
Time Frame: Time in recovery room, approximately 60-90 minutes.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 16
mg/kg | 0.07 (0.05) | 0.03 (0.04)

3. Secondary Outcome: Assessment of First Pain Score on Arrival to Recovery Room.
Description: Pain scores will be assessed using the Faces-Legs-Activity-Cry-Consolibility (FLACC) scale for children ≤ 7 years old. The FLACC scale is from 0-10 (0=no pain, 10=worst pain). The scale is composed of five subscales (Faces = facial expression; Legs = lower extremity movement; Activity = degree of movement; Cry = how upset the child is; Consolibity = how easy the child can be consoled). Eacg subscale is rated 0 to 2 (0 = rated as comfortable, no or minimal discomfort for that subscale; 2 = rated as uncomfortable, in pain according to that subscale). The subscales are summed to give a composite score out of 10. Pain scores will be assessed at admission to the recovery room.
Time Frame: On arrival to recovery room.
Measure: Mean (Standard Deviation); unit: units on FLACC pain scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 16
units on FLACC pain scale | 5 (5) | 2 (3)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No